CLINICAL TRIAL: NCT01204164
Title: Phase 1 Dose-Escalation and Pharmacokinetic Study of TG02 Citrate in Patients With Advanced Hematological Malignancies
Brief Title: Phase 1 Study of TG02 Citrate in Patients With Advanced Hematological Malignancies
Acronym: TG02-101
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tragara Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TG02-101
Record Dates: First submitted 2010-09-14; First posted 2010-09-17 (Estimated); Last update posted 2016-05-06 (Estimated); Status verified 2016-05

CONDITIONS: AML; ALL; Blast Crisis; MDS; Multiple Myeloma
Keywords: AML; ALL; MDS; CML in blast crisis; Multiple Myeloma; Carfilzomib refractory
MeSH Terms: conditions — Blast Crisis; Multiple Myeloma | interventions — carfilzomib; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- TG02 in AL (Experimental): Single agent TG02 citrate in acute leukemia patients
  Interventions: Drug: TG02 citrate
- TG02 in MM (Experimental): Single Agent TG02 citrate in multiple myeloma patients
  Interventions: Drug: TG02 citrate
- TG02 + CFZ in MM (Experimental): TG02 in combination with carfilzomib and dexamethasone in multiple myeloma patients
  Interventions: Drug: TG02 citrate; Drug: Carfilzomib
- TG02 + CFZ + DEX in CFZ refractory MM (Experimental): TG02 in combination with carfilzomib and dexamethasone in carfilzomib refractory multiple myeloma patients
  Interventions: Drug: TG02 citrate; Drug: Carfilzomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: TG02 citrate — TG02 citrate capsules given orally.
  Other Names: No other names.
Drug: Carfilzomib — Carfilzomib per PI
  Other Names: Kyprolis
  Arms: TG02 + CFZ + DEX in CFZ refractory MM; TG02 + CFZ in MM
Drug: Dexamethasone — Dexamethasone (Oral or IV)
  Other Names: Ozurdex, Maxidex, Decadron, Baycadron
  Arms: TG02 + CFZ + DEX in CFZ refractory MM

SUMMARY:
This is a multicenter, open-label, dose escalation Phase 1 study.

DETAILED DESCRIPTION:
This is a multicenter, open-label, dose escalation, Phase 1/1b study.

For Parts 1, 2, and 3 of the study, the primary objective is to determine the highest dose of TG02 citrate that can safely be given to patients with different types of hematological malignancy.

For Part 4, the primary objective is to evaluate the safety and tolerability of once-weekly dosing at the maximum-tolerated dose/ Recommended Phase 2 Dose of TG02 in combination with carfilzomib.

This study consists of four parts:

* Part 1: single agent TG02 in acute leukemia patients
* Part 2: single agent TG02 in multiple myeloma patients
* Part 3: TG02 in combination with carfilzomib in multiple myeloma patients
* Part 4: TG02 in combination with carfilzomib in carfilzomib refractory multiple myeloma patients.

ELIGIBILITY:
Part 1 Inclusion Criteria:

* Relapsed AML, ALL, CML in blast crisis, or MDS
* 65+ yrs with AML not eligible for standard frontline chemo
* Interval from prior treatment to time of study drug at least 5 half-lives for cytotoxic/ noncytotoxic agents.
* Persistent clinically significant toxicities from prior chemo ≤ Grd 1
* ECOG PS 0-2
* Lab values:

  * Cr ≤ 2X ULN
  * ALT and/or AST ≤2.5 X ULN
  * Total bilirubin ≤1.5 X ULN unless considered due to Gilbert's syndrome
* Negative pregnancy test
* Can take oral med

Part 2 Inclusion Criteria:

* Relapsed multiple myeloma. At least ≥1 line of therapy and progressed after ≥1 prior therapy
* Measurable disease defined as at least one of the following:

  * Serum M ≥500 mg/dL
  * Urine M ≥200 mg per 24hr
  * Involved FLC ≥10 mg/dL and abnormal FLC ratio in serum (<0.26 or >1.65)
  * Measurable soft tissue plasmacytoma
* Persistent clinically significant toxicities from prior chemo ≤ Grd 1
* ECOG PS 0-2
* Lab values:

  * ANC of >1000/mm3
  * Platelets ≥50,000/mm3
  * Cr ≤2X the ULN
  * ALT and/or AST ≤2.5X ULN
  * Total bilirubin ≤1.5X ULN, unless considered due to Gilbert's syndrome
* Negative pregnancy test
* Can take oral med

Part 3 Inclusion Criteria:

* Measurable disease defined as at least one of the following:

  * Serum M ≥500 mg/dL
  * Urine M protein ≥200 mg per 24hr
  * Involved FLC level ≥10 mg/dL and abnormal FLC ratio in serum (<0.26 or >1.65)
* Meet at least one of the criteria below:

  * a. ≥2 prior therapies including proteasome inhibitor and immunomodulatory agent (IMiD)
  * b. ≥1 prior therapy and one of the following abnormalities: 17p del, p53, 1q amp, 1p del, t(4;14)
* Interval from prior treatment to time of study drug at least 5 half-lives or 3 wks, which ever is shorter, for noncytotoxic agents
* Persistent clinically significant toxicities from prior chemo ≤ Grd 1 or Grd 2 neuropathy without pain
* ECOG PS 0-2
* Lab values:

  * ANC of >1000/mm3 independent of G-CSF
  * Platelets ≥50,000/mm3 independent of transfusion
  * MDRD calculated or measured CrCl of ≥30 mL/min
  * ALT and/or AST ≤3X ULN
  * Total bilirubin ≤2X ULN, unless considered due to Gilbert's syndrome
* Negative pregnancy test
* Can take oral med

Part 4 Inclusion Criteria:

* Measurable disease defined as at least one of the following:

  * Serum M ≥500 mg/dL
  * Urine M protein ≥200 mg per 24hr
  * Involved FLC level ≥10 mg/dL and an abnormal FLC ratio in serum (<0.26 or >1.65)
* Received prior therapies including:

  * a. bortezomib
  * b. an IMiD
  * c. carfilzomib. Demonstrated disease progression on or within 60d of completion of carfilzomib therapy
* Interval from prior treatment to time of study drug at least 5 half-lives or 3 wks, which ever is shorter, for noncytotoxic agents.
* Persistent clinically significant toxicities from prior chemo ≤ Grd 1, or Grd 2 neuropathy without pain.
* ECOG PS 0-2
* Lab values:

  * ANC of >1000/mm3 independent of G-CSF
  * Platelets ≥50,000/mm3 independent of transfusion
  * MDRD calculated or measured CrCl of ≥30 mL/min
  * ALT and/or AST ≤3X ULN
  * Total bilirubin ≤2X ULN, unless considered due to Gilbert's syndrome
* Negative pregnancy test
* Can take oral med

Parts 1 and 2 Exclusion Criteria:

* Previous allogenic hematopoietic transplant within 90 d
* Concurrent severe or uncontrolled medical disease that would compromise the safety or compromise the ability of the patient to complete the study
* Prolonged QTC interval >450ms
* Symptomatic CNS metastases
* Known HIV or AIDS
* Actively treated for a second malignancy
* Pregnant or nursing women

Part 3 Exclusion Criteria:

* Multiple myeloma of IgM subtype, POEMS, plasma cell leukemia
* Corticosteroids discontinued ≥7 days of initiating therapy
* Previous chemo within 2 wks
* Hx of ventricular arrhythmia or symptomatic conduction abnormality within 12m
* CHF, symptomatic ischemia, conduction abnormalities uncontrolled by conventional intervention, myocardial infarction within 6m
* Prolonged QTc interval (males >450ms, females >470ms)
* Previous allogeneic hematopoietic transplant within 90 days of study enrollment, Active GVHD requiring treatment.
* Concurrent severe or uncontrolled medical disease that would compromise the safety or compromise the ability of the patient to complete the study
* Symptomatic CNS metastases
* Known HIV or AIDS
* Prior or 2nd malignancy, except non-melanoma skin cancer, completely resected cervical or prostate cancer (with PSA of less than or equal to 0.1 ng/ml), or other cancer for which the subject has received curative therapy at least 3 yrs prior to study entry
* Treatment-related MDS
* Significant neuropathy (Grd 3-4 or Grd 2 with pain) at the time of 1st dose
* Primary AL amyloidosis
* Pleural effusions requiring thoracentesis or ascites requiring paracentesis
* Pregnant or nursing women

Part 4 Exclusion Criteria:

* Multiple myeloma of IgM subtype, POEMS, plasma cell leukemia
* Previous chemo within 2 wks
* Hx ventricular arrhythmia or symptomatic conduction abnormality within 12m
* CHF, symptomatic ischemia, conduction abnormalities uncontrolled by conventional intervention, and myocardial infarction within 6m
* Prolonged QTc interval (males >450ms, females >470ms)
* Previous allogeneic hematopoietic transplant within 90 days. Active GVHD requiring treatment
* Concurrent severe or uncontrolled medical disease that would compromise the safety or compromise the ability of the patient to complete study
* Symptomatic CNS metastases
* Known HIV or AIDS
* Prior or 2nd malignancy, except non-melanoma skin cancer, completely resected cervical or prostate cancer (with PSA of less than or equal to 0.1 ng/ml), or other cancer for which the subject has received curative therapy at least 3 yrs prior to study entry
* Treatment-related MDS
* Significant neuropathy (Grd 3-4 or Grd 2 with pain) at the time of 1st dose
* Primary AL amyloidosis
* Pleural effusions requiring thoracentesis or ascites requiring paracentesis
* Pregnant or nursing women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2010-08; Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | 28 days
  Maximum Tolerated Dose refers to the highest dose of TG02 administered that will produce the desired effect without unacceptable toxicity.

SECONDARY OUTCOMES:
Safety | 28 days
  Safety data will include vital signs, ECGs, PE findings, clinical laboratory parameters, ECOG PS, AEs/SAEs and concomitant medications.
Pharmacokinetics of TG02 | 28 days
  Plasma will be analyzed to determine TG02 concentration.
Clinical Benefit Response | 28 days
  Clinical Benefit Response is defined as the sum of all response categories for Overall Response Rate (ORR is defined as the sum of patients with sCR, CR, VGPR and PR) plus minimal response (MR).
Overall Response Rate | 28 days
  Overall Response Rate is defined as the sum of patients with sCR, CR, VGPR and PR.
Progression-Free Survival | 28 days
  Progression-Free Survival is the time to disease progression or death, which is measured from the date of first study drug administration until the first date that recurrent or progressive disease is objectively documented or the date of death.
Overall Survival | 28 days
  Overall Survival is time to death, which is measured from the date of first study drug administration until the date of death.
Duration of Response | 28 days
  Duration of Response is the duration from first observation of response to the first documentation of disease progression, with deaths from causes other than disease progression censored. For the purposes of the calculation of the DOR, the date at which the response status was first observed rather than the date of confirmation is used as the start date.
Pharmacodynamics | 28 days
  Pharmacodynamic sampling may include whole blood and bone marrow at baseline and post-treatment for pathway determination if available.

CONTACTS AND LOCATIONS:
Overall Officials: T Parrott, Study Director — Tragara Pharmaceuticals
Locations (9):
- United States (9):
  - RMCC, Denver, Colorado
  - Emory, Atlanta, Georgia
  - Rush, Chicago, Illinois
  - IU, Indianapolis, Indiana
  - HUMC, Hackensack, New Jersey
  - Cornell, New York, New York
  - OSU, Columbus, Ohio
  - SCRI, Nashville, Tennessee
  - MDACC, Houston, Texas